CLINICAL TRIAL: NCT04594408
Title: The Use of Tranexamic Acid in Irrigation Fluid to Improve Arthroscopic Visualization in Shoulder Surgery: A Randomized Controlled Trial
Brief Title: Tranexamic Acid to Improve Arthroscopic Visualization in Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA2018-001
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Tears; Subacromial Impingement; Subacromial Impingement Syndrome
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome | interventions — Epinephrine; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons are blinded to group allocation as all IV bags will have labels appearing identical when turned away from the surgeon. Anesthetists are told not to reveal allocation to the surgeon as well. And patients will not be informed of their allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- No epinephrine or TXA (No Intervention): No intervention given.
- Epinephrine in irrigation fluid (Active Comparator): Epinephrine intervention used.
  Interventions: Drug: Epinephrine
- Intravenous TXA (Experimental): Tranexamic acid intervention used.
  Interventions: Drug: Tranexamic acid
- Epinephrine and TXA (Experimental): Epinephrine and tranexamic acid intervention used.
  Interventions: Drug: Epinephrine and Tranexamic Acid

INTERVENTIONS:
Drug: Epinephrine — 1 mL of 1:1000 mixed into irrigation bag.
  Other Names: Epi
  Arms: Epinephrine in irrigation fluid
Drug: Tranexamic acid — 1 g IV x 1 dose to be administered intraoperatively.
  Other Names: TXA
  Arms: Intravenous TXA
Drug: Epinephrine and Tranexamic Acid — 1 mL of 1:1000 epinephrine mixed into irrigation bag, and 1 g tranexamic acid x 1 dose to be administered intraoperatively.
  Other Names: TXA, Epi
  Arms: Epinephrine and TXA

SUMMARY:
The purpose of this study is to determine if intravenous TXA is a safe alternative to epinephrine in improving arthroscopic shoulder visualization.

Primary Objectives

1. Determine that patients given intravenous tranexamic acid improves surgeon-rated visualization compared to placebo.
2. Determine that intravenous tranexamic acid is a safe alternative to epinephrine mixed irrigation fluid to improve arthroscopic shoulder visualization

DETAILED DESCRIPTION:
In the last twenty years, the use of arthroscopy to surgically manage shoulder pathologies has expanded in its indications. The interplay between increased indications, surgeon experience, and improvements in equipment have all propelled arthroscopic shoulder surgery to preferred treatment in managing instability, rotator cuff, and impingement pathology. Obtaining adequate visual clarity is paramount to performing the procedures safely, efficiently, and effectively.

A variety of methods have been employed to improve visualization. This includes tighter control of blood pressure, regional anesthetic, pressure controlled irrigation system, sealed cannulas, electrocautery devices, and injecting epinephrine into irrigation fluid. The use of epinephrine in irrigation fluid has been studied in literature. The results of a few randomized controlled trials demonstrate that the vasoconstrictive properties of epinephrine decrease blood flow and consequently, improves surgeon visualization. However, there has been reports of ventricular tachycardia, lethal arrhythmias, and epinephrine induced pulmonary edema in literature that suggests that the addition of epinephrine in irrigation fluid may have caused these adverse events. Therefore, it is important to examine other alternatives, such as TXA, that can decrease bleeding and improve visualization without potential detrimental effects.

This trial will be conducted in compliance with the protocol, GCP, and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand patient consent form and give informed consent
* Rotator cuff pathology or impingement that have clinical indications for shoulder arthroscopy surgery (either rotator cuff repair or subacromial decompression

Exclusion Criteria:

* Have an active thromboembolic event
* Allergies or hypersensitivies to TXA or any of the ingredients
* Have a seizure disorder
* On hormonal contraceptives
* Pregnant
* History of venous thromboembolism in the previous 12 months, or requiring lifelong anticoagulation related to previous VTE. VTE is defined as a cerebrovascular event (stroke, transient ischemic attack, deep vein thrombosis, and pulmonary embolism or with a history of hypercoagulable disorders (i.e. Factor V Lieden, antiphospholipid antibody)
* Acquired disturbances of colour vision
* Hematuria with renal cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Visualization Quality Scale | Intra-operative
  Surgeons are asked every 15 minutes to report on the quality of visualization based on a 4-point scale. Minimum value is 0, maximum value is 3 with the higher value reflecting improved visualization

SECONDARY OUTCOMES:
Patient Log Book for Pain and Medications | Day of surgery - post-operative day 14
  Patients are sent home from surgery with a log book to track the level of pain they are experiencing as well as the medications that they take.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Old, MD, FRCSC, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Jensen KH, Werther K, Stryger V, Schultz K, Falkenberg B. Arthroscopic shoulder surgery with epinephrine saline irrigation. Arthroscopy. 2001 Jul;17(6):578-81. doi: 10.1053/jars.2001.23590. PMID 11447543
- [Background] Morrison DS, Schaefer RK, Friedman RL. The relationship between subacromial space pressure, blood pressure, and visual clarity during arthroscopic subacromial decompression. Arthroscopy. 1995 Oct;11(5):557-60. doi: 10.1016/0749-8063(95)90131-0. PMID 8534296
- [Background] Ogilvie-Harris DJ, Weisleder L. Fluid pump systems for arthroscopy: a comparison of pressure control versus pressure and flow control. Arthroscopy. 1995 Oct;11(5):591-5. doi: 10.1016/0749-8063(95)90137-x. PMID 8534302
- [Background] Avery DM 3rd, Gibson BW, Carolan GF. Surgeon-rated visualization in shoulder arthroscopy: a randomized blinded controlled trial comparing irrigation fluid with and without epinephrine. Arthroscopy. 2015 Jan;31(1):12-8. doi: 10.1016/j.arthro.2014.08.010. Epub 2014 Nov 6. PMID 25442659
- [Background] van Montfoort DO, van Kampen PM, Huijsmans PE. Epinephrine Diluted Saline-Irrigation Fluid in Arthroscopic Shoulder Surgery: A Significant Improvement of Clarity of Visual Field and Shortening of Total Operation Time. A Randomized Controlled Trial. Arthroscopy. 2016 Mar;32(3):436-44. doi: 10.1016/j.arthro.2015.08.027. PMID 26524933
- [Background] Mazzocca AD, Meneghini RM, Chhablani R, Badrinath SK, Cole BJ, Bush-Joseph CA. Epinephrine-induced pulmonary edema during arthroscopic knee surgery. A case report. J Bone Joint Surg Am. 2003 May;85(5):913-5. doi: 10.2106/00004623-200305000-00023. No abstract available. PMID 12728044
- [Background] Cho SH, Yi JW, Kwack YH, Park SW, Kim MK, Rhee YG. Ventricular tachycardia during arthroscopic shoulder surgery: a report of two cases. Arch Orthop Trauma Surg. 2010 Mar;130(3):353-6. doi: 10.1007/s00402-009-0820-1. Epub 2009 Jan 29. PMID 19184069
- [Background] Karns JL. Epinephrine-induced potentially lethal arrhythmia during arthroscopic shoulder surgery: a case report. AANA J. 1999 Oct;67(5):419-21. PMID 10876433
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Benoni G, Fredin H. Fibrinolytic inhibition with tranexamic acid reduces blood loss and blood transfusion after knee arthroplasty: a prospective, randomised, double-blind study of 86 patients. J Bone Joint Surg Br. 1996 May;78(3):434-40. PMID 8636182
- [Background] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147
- [Background] Zhou XD, Tao LJ, Li J, Wu LD. Do we really need tranexamic acid in total hip arthroplasty? A meta-analysis of nineteen randomized controlled trials. Arch Orthop Trauma Surg. 2013 Jul;133(7):1017-27. doi: 10.1007/s00402-013-1761-2. Epub 2013 Apr 25. PMID 23615973
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Huang F, Wu D, Ma G, Yin Z, Wang Q. The use of tranexamic acid to reduce blood loss and transfusion in major orthopedic surgery: a meta-analysis. J Surg Res. 2014 Jan;186(1):318-27. doi: 10.1016/j.jss.2013.08.020. Epub 2013 Sep 13. PMID 24075404
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Tan J, Chen H, Liu Q, Chen C, Huang W. A meta-analysis of the effectiveness and safety of using tranexamic acid in primary unilateral total knee arthroplasty. J Surg Res. 2013 Oct;184(2):880-7. doi: 10.1016/j.jss.2013.03.099. Epub 2013 Apr 25. PMID 23643299